CLINICAL TRIAL: NCT01992640
Title: Recovery After Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anne Kathrine Staehr-Rye, M.D., Herlev Hospital
Other Study IDs: 11-2013
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
During laparoscopic surgery, muscle relaxants are often administrated in order to ensure acceptable surgical conditions. These drugs bind to receptors in the neuromuscular junction.

The degree of muscle relaxation is monitored by use of an acceleromyography and at the end of surgery another drug - Neostigmine- is given to reverse the muscle relaxation. However,there may still be a blockade of up to 70% of the receptors.

This partial muscle relaxation may result in muscle weakness, reduced balance and prolonged hospitalization.

This study will describe changes in balance and subjective muscle weakness after laparoscopic surgery.

The primary hypothesis is that sway area is increased 30 min after extubation compared to the preoperative value.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Same-day gynaecological laparoscopic surgery
* Informed consent

Exclusion Criteria:

* Body mass index above 30 kg/m2
* Insufficient renal function
* Liver insufficience
* Neuromuscular monitoring not possible
* Known allergy towards medicine used in the protocol
* Daily use of opioids
* Known disease which can interfere with the balance
* Pregnant/lactating
* Cannot read or understand danish
* Fast-track intubation with use of succinylcholine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients scheduled for laparoscopic surgery at Herlev Hospital and expected discharge on the same day as surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in postural sway area 30 min after extubation (closed eyes) | Preoperatively and 30 min after extubation

SECONDARY OUTCOMES:
Change in sway area when ready to be discharge form the postoperative care unit (PACU)(closed eyes) | Preoperatively and at discharge from the PACU. An expected duration of 2 hours after surgery
change in sway area 30 min after extubation (open eyes) | Preoperatively and 30 min after extubation
Change in sway area when ready to be discharged from the PACU (open eyes) | Preoperatively and when ready to be discharged from the PACU. An expected average of 2 hours after surgery
Change in sway velocity 30 min after extubation (closed eyes) | Preoperatively and 30 min after extubation
Change in sway velocity 30 min after extubation (open eyes) | Preoperatively and 30 min after extubation
Change in sway velocity when ready to be discharged from the PACU (closed eyes) | Preoperatively and when ready to be discharged from the PACU. An expected duration of 2 hours after surgery
Change in sway velocity when ready to be discharged from the PACU (open eyes) | Preoperatively and when ready to be discharged from the PACU. An expected duration of 2 hours after surgery
Change in mean sway 30 min after extubation (closed eyes) | Preoperatively and 30 min after extubation
Change in mean sway 30 min after extubation (open eyes) | Preoperatively and 30 min after extubation
Change in mean sway when ready to discharge from the PACU (closed eyes) | Preoperatively and when ready to be discharged from the PACU. An expected duration of 2 hours after surgery.
Change in mean sway when ready to be discharged from the PACU (open eyes) | Preoperatively and when ready to be discharged from the PACU. An expected duration of 2 hours after surgery
Change in subjective balance 30 min after extubation | Preoperatively and 30 min after extubation
Change in subjective balance when ready to be discharged from the PACU | Preoperatively and when ready to be discharged from the PACU. An expected duration of 2 hours after surgery
Change in muscle weakness 30 min after extubation | Preoperatively and 30 min after extubation
Change in muscle weakness when ready to be discharged from the PACU | preoperatively and when ready to be discharge from the PACU. An expected duration of 2 hours
Incidence of critical respiratory events from extubation until discharge from the PACU | From extubation until discharge from the PACU (approximately 2 hours)
Duration of stay at the PACU | The patients will be followed from extubation until leaving the PACU. An expected average duration of 2 hours
Duration of postoperative hospitalization | The patient will be followed from extubation until discharge from hospital. An expected average duration of 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Staehr-Rye, M.D., Principal Investigator — Dept. of Anesthesiology, Herlev Hospital; Mona R Gätke, M.D.; Ph.D., Study Chair — Dept. of Anesthesiology, Herlev Hospital
Locations (1):
- Dept. of Anesthesiology, University of Copenhagen, Herlev Hospital, Herlev, Denmark